CLINICAL TRIAL: NCT04058483
Title: A Randomized Trial Validating the New Remote Hypnotic Induction Profile (rHIP) Against the Existing Hypnotic Induction Profile (HIP)
Brief Title: Validating the New Remote Hypnotic Induction Profile (rHIP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jessie Kittle, Assitant Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 51970
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Testing the Hypnotizability of Healthy Volunteers
Keywords: hypnosis; hypnotizability; validation; remote; Hypnotic Induction Profile

STUDY DESIGN:
Intervention Model Description: Participants are randomized to first undergo phone-administered testing vs. in-person testing.
Who Masked: Participant, Investigator
Masking Description: Participants not told their hypnotizability score from the first exam prior to completing the second exam.
  Study personnel performing the second hypnotizability test are masked to the first hypnotizability score. Two separate investigators will test each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIP First (Active Comparator): Participants randomized to perform the in-person hypnotizability test first. This will be followed within 1 week with the by-phone rHIP test performed by a second, randomly-assigned investigator.
  Interventions: Other: Hypnotizability testing
- rHIP First (Active Comparator): Participants randomized to perform the by-phone hypnotizability test first. This will be followed within 1 week with the in-peron HIP test performed by a second, randomly-assigned investigator.
  Interventions: Other: Hypnotizability testing

INTERVENTIONS:
Other: Hypnotizability testing — Hypnotizability testing in-person vs. by phone. All participants will complete both conditions.

SUMMARY:
The purpose of the study is to determine if hypnotizability can be reliably tested over the phone, without having to see or touch a patient. The scores from a new test for hypnotizability by phone will be compared to the scores from a standard in-person test, to make sure the results are similar.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old.
* Able to schedule a 15 minute in-person and phone appointment within a week of each other, during the study period.

Exclusion Criteria:

* Severe psychiatric or structural brain disease (ie. psychosis, stroke with functional impairment, dementia)
* Has had prior hypnotizability testing using the HIP or enrolled in another hypnosis-related trial.
* hearing impairment that would preclude phone interviewing
* non-English speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2019-10-14 (Actual); Study Completion 2019-10-14 (Actual)

PRIMARY OUTCOMES:
Reliability of HIP and rHIP test scores | Through study completion, approximately 2 months.
  Calculate the correlation between the HIP and rHIP

SECONDARY OUTCOMES:
Hypnotizability and DES | Administered upon enrollment, prior to first hypnotizability test
  Investigate any correlation between hypnotizability scores and the Dissociative Experiences Scale
Hypnotizability and Tellegen | Administered upon enrollment, prior to first hypnotizability test
  Investigate any correlation between hypnotizability scores and the Tellegen Absorption Scale
Complications with phone-administered test | Through study completion, approximately 2 months.
  Researchers will recored the % of participants who reported technical or practical difficulties with the phone-administered test including difficulty hearing, understanding the instructions, getting interrupted during the test, or others.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University/Stanford Healthcare, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Please email PI for data if interested.

REFERENCES:
- [Derived] Kittle J, Zhao E, Stimpson K, Weng Y, Spiegel D. Testing Hypnotizability by Phone: Development and Validation of the Remote Hypnotic Induction Profile (rHIP). Int J Clin Exp Hypn. 2021 Jan-Mar;69(1):94-111. doi: 10.1080/00207144.2021.1827937. PMID 33513064